CLINICAL TRIAL: NCT00974376
Title: Gabapentin Treatment of Cannabis Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Scripps Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Barbara J. Mason, PI, The Scripps Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA026758; 5R01DA026758-05 (NIH)
Record Dates: First submitted 2009-09-01; First posted 2009-09-10 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Cannabis Dependence; Cannabis Withdrawal; Cognitive Deficits
Keywords: Cannabis Treatment; Cannabis Use; Cannabis Dependence; Executive Functioning; Cognitive Deficits
MeSH Terms: conditions — Marijuana Abuse; Cognition Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin 1200mg/day (Experimental): 1200mg/day of gabapentin for 12 weeks given in conjunction with 12 weeks of manual-guided behavioral counseling.
  Interventions: Drug: gabapentin 1200mg/day; Behavioral: Manual-guided behavioral counseling
- Placebo (Placebo Comparator): 1200mg/day of placebo for 12 weeks given in conjunction with 12 weeks of manual-guided behavioral counseling.
  Interventions: Drug: Placebo; Behavioral: Manual-guided behavioral counseling

INTERVENTIONS:
Drug: gabapentin 1200mg/day — gabapentin 1200mg/day for 12 weeks
  Other Names: Neurontin
  Arms: Gabapentin 1200mg/day
Drug: Placebo — 1200mg/day of placebo for 12 weeks
  Arms: Placebo
Behavioral: Manual-guided behavioral counseling — Standardized manual-guided behavioral counseling performed 1 time per week for 12 weeks in conjunction with study drug or placebo.
  Other Names: Manual-guided therapy

SUMMARY:
This is a clinical study to evaluate the efficacy of the medication gabapentin in treating persons with cannabis dependence.

DETAILED DESCRIPTION:
This is a 12-week, double blind, placebo controlled study to evaluate the efficacy of gabapentin in treating outpatients with cannabis dependence. After an initial phone screen, a comprehensive screening visit is scheduled to determine eligibility. Upon enrollment, counseling, medication dispensation and research assessments occur 1 time per week for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females from 18-65 years of age
* Meets DSM IV criteria for current cannabis dependence
* Seeking research-based outpatient treatment for cannabis dependence that involves daily medication
* Smoked MJ daily at least 25 days per month during the 90 days prior to randomization
* At least a 2-year history of regular MJ use

Exclusion Criteria:

* Abstinent from cannabis more than 2 days at the time of randomization
* Active suicidal ideation
* Currently meets DSM IV criteria for abuse or dependence on other substances, or has urine drug screen positive for substances, other than cannabis or nicotine
* Significant medical disorders that will increase potential risk or interfere with study participation,
* Sexually active female participants with childbearing potential who are pregnant, nursing or refuse to use a reliable method of birth control
* Meets DSM IV criteria for a major AXIS I disorder other than cannabis and nicotine dependence,
* Inability to understand and/or comply with the provisions of the protocol and consent form
* Treatment with an investigational drug during the previous month
* Sensitivity to study drug as evidenced by adverse drug experiences with gabapentin or its ingredients
* Ongoing treatment with medications that may affect study outcomes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-11-04 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Mason, Ph.D., Principal Investigator — The Scripps Research Institute
Locations (1):
- The Scripps Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — http://alcoholismmarijuanatreatment.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin 1200mg/Day: 1200mg/day of gabapentin given in conjunction with standardized manual-guided behavioral counseling.
- Placebo: Matched placebo given in conjunction with standardized manual-guided behavioral counseling.
Period: Overall Study
Arm/Group | Gabapentin 1200mg/Day | Placebo
Started | 75 | 75
Completed | 41 | 42
Not Completed | 34 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin 1200mg/Day | Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.99 (10.68) | 34.53 (11.99) | 34.76 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 52 | 48 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Negative Urinary Drug Screens (UDS) for Cannabis at 12 Weeks Following Administration of Gabapentin or Placebo During the Double Blind Period
Description: Express Results Integrated Multi-Drug Screen Cups were used to obtain a semi-quantitative urine drug screen for delta-9-THC. Submitted UDS would yield a positive result when the concentration of THC-COOH in urine exceeded 50 ng/mL. Specimens were collected weekly. Two analytical approaches were used: one where any missed UDS test was assumed positive (i.e intent-to-treat (ITT)) and another where missed UDS were considered missing at random (MAR).
Time Frame: 12 weeks
Population: Two participants in the gabapentin group and one in the placebo group were lost to follow up after randomization and did not submit any UDS for testing while on study. Two participants in the placebo group withdrew from the study at the week 1 visit, and thus did not submit any UDS for testing while on study.
Measure: Mean (Standard Deviation); unit: percentage of negative UDS
Arm/Group | Gabapentin 1200mg/Day | Placebo
Number analyzed (Participants) | 75 | 75
percentage of negative UDS
  % Negative UDS ITT | 11.22 (21.77) | 8.00 (19.83)
  % Negative UDS Observed: number analyzed (Participants) | 73 | 72
  % Negative UDS Observed | 12.48 (23.82) | 9.93 (24.03)

ADVERSE EVENTS:
Arm/Group | Gabapentin 1200mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 0/150 | 1/150
Other Adverse Events (participants affected / at risk) | 40/75 | 50/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin 1200mg/Day (N=150) | Placebo (N=150)
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin 1200mg/Day (N=75) | Placebo (N=75)
Diarrhoea (Gastrointestinal disorders) | 5 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 8 | 8
Vomiting (Gastrointestinal disorders) | 4 | 2
Fatigue (General disorders) | 10 | 3
Nasopharyngitis (Infections and infestations) | 14 | 19
Urinary tract infection (Infections and infestations) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Dizziness (Nervous system disorders) | 6 | 7
Headache (Nervous system disorders) | 11 | 15
Somnolence (Nervous system disorders) | 7 | 5
Insomnia (Psychiatric disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No